CLINICAL TRIAL: NCT00117624
Title: A Randomized, Double-Blind, Study of Front-Loading Darbepoetin Alfa Compared With Standard Weekly Administration for the Treatment of Anemia in Subjects With a Non-Myeloid Malignancy and Receiving Multicycle Chemotherapy
Brief Title: A Study of Darbepoetin Alfa for the Treatment of Anemia in Subjects With a Non-Myeloid Malignancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20020118
Record Dates: First submitted 2005-06-30; First posted 2005-07-08 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Anemia
Keywords: Non-myeloid malignancy; Darbepoetin alfa; Clinical Trial
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa

SUMMARY:
The purpose of this study is to compare the efficacy of darbepoetin alfa administered using a front-loading approach with subjects receiving standard weekly dosing in the treatment of anemia in subjects with a non-myeloid malignancy and receiving multicycle chemotherapy.

ELIGIBILITY:
Inclusion Criteria: - Non-myeloid malignancy - At least 12 additional weeks of cyclic cytotoxic chemotherapy anticipated regardless of schedule - ECOG 0-2 - Cancer and/or chemotherapy-associated anemia Exclusion Criteria: - Known history of seizure disorder - Known primary hematologic disorder, which could cause anemia, other than a non-myeloid malignancy - Unstable or uncontrolled disease/condition, related to or affecting cardiac function - Clinically significant inflammatory disease - Inadequate renal and/or liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-12; Study Completion 2003-12

PRIMARY OUTCOMES:
RBC transfusion during the treatment phase

SECONDARY OUTCOMES:
The time to hemoglobin response during the treatment phase
The FACT-Fatigue score profile over time
The change in hemoglobin
Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Kotasek D, Canon JL, Mateos MV, Hedenus M, Rossi G, Taylor K. A randomized, controlled trial comparing darbepoetin alfa correction/maintenance dosing with weekly dosing for treating chemotherapy-induced anemia. Curr Med Res Opin. 2007 Jun;23(6):1387-401. doi: 10.1185/030079907X188053. Epub 2007 May 8. PMID 17559735
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com